CLINICAL TRIAL: NCT04681664
Title: Development of Methods and Algorithms to Design Diets Based on Gut Microbiome Analysis
Brief Title: Gut Microbiome Based Analysis of High Protein High Fat Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center of Food and Fermentation Technologies (Other)
Collaborators: National Institute for Health Development, Estonia (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NSP67
Record Dates: First submitted 2020-11-30; First posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Obesity
Keywords: microbiome; ribosomal sequencing; obesity; bifidobacteria; Collinsella
MeSH Terms: conditions — Obesity | interventions — Diet, High-Fat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 50 % fat diet (Experimental): In the high fat group the subjects were assigned to the diet containing in average 50 % fat, 25 % proteins and 25 % carbohydrates for four weeks.
  Interventions: Other: High fat diet

INTERVENTIONS:
Other: High fat diet — 50 % fat

SUMMARY:
The aim of this study was to determine body mass reduction and microbiota composition change after the weight loss diet (50 % fat, 25 % proteins and 25 % carbohydrates).

DETAILED DESCRIPTION:
For high fat group a total of 19 overweight/obese participants (14 females, 5 males, aged 25 to 43) with BMI of 28.9-44.4 kg/m2 were assigned to low-calorie low-carbohydrate high-fat weight loss diet for 4 weeks.

As a control group, 58 subjects (39 females, 20 males, aged 24 to 55 years) were recruited and divided into 3 groups based on BMI: 18-25, 25-30, 30-39 kg/m2 (N=33, N=16, N=9, respectively).

Inclusion criteria for participants included no previous history of gastrointestinal (GI) disease, no reported antibiotic use in preceding 3 months, or taking any medication known to alter bowel motility, no history of food allergies and not taking medications.

Before the study all participants were informed about the study and participants were signed a written consent.

At day 0 baseline samples and data were collected (faecal sample, Bristol score and bowel habits, food diary about the period of at least three days before faecal sampling, body weight). After collection of baseline samples subjects in the high fat group started diet plan for 4 weeks while control group contiunued their habitual diet. After the 4 week intervention period samples and data were collected again (faecal sample, Bristol score and bowel habits, food diary about the period of at least three days before faecal sampling, body weight).

ELIGIBILITY:
Inclusion Criteria for obese group:

* BMI > 30 g/m2

Exclusion Criteria:

* antibiotic treatment within last three months;
* food restrictions due to allergies, any kind of food intolerance, veganism/vegetarianism or other extremes in food consumption practices;
* chronic illnesses;
* current pregnancy or breastfeeding
* travel to subtropical or tropical regions within one month before the study.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Decrease of body weight during 4 weeks high fat diet | Baseline and after 4 weeks
  Body weight was measured by calibrated scale before the study (baseline) and after the diet intervention (4 week)
Reduction of inflammation related bacteria in faecal microbiota | 4 weeks
  Bacterial composition was measured by 16S ribosomal sequencing at baseline and after the 4 weeks diet. The relative change of each bacterial taxon was calculated based on the abundance of the given bacteria at baseline and after 4 weeks high fat diet.

CONTACTS AND LOCATIONS:
Locations (1):
- Center of Food and Fermentation Technologies, Tallinn, Harju, Estonia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol: Study protocol (2016-10-25): https://cdn.clinicaltrials.gov/large-docs/64/NCT04681664/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-25): https://cdn.clinicaltrials.gov/large-docs/64/NCT04681664/SAP_001.pdf
  • Informed Consent Form (2016-10-25): https://cdn.clinicaltrials.gov/large-docs/64/NCT04681664/ICF_002.pdf